CLINICAL TRIAL: NCT01937481
Title: A Longitudinal Study to Assess if the Effectiveness of a Preschool Nutrition and Physical Activity Program is Sustained in Elementary School
Brief Title: The Colorado LEAP Study: A Socioecological Approach to Obesity Prevention in Early Childhood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency); University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: USDA NIFA 2010-85215-20648
Record Dates: First submitted 2013-08-28; First posted 2013-09-09 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Childhood Obesity
Keywords: Child, Preschool; Parents; Family; Obesity; Overweight; Diet; Overnutrition; Motor Activity; Child Care; Schools
MeSH Terms: conditions — Pediatric Obesity; Obesity; Overweight; Overnutrition; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutrition and Physical Activity (Experimental): The Food Friends programs
  Interventions: Behavioral: The Food Friends
- Control (No Intervention): Control group

INTERVENTIONS:
Behavioral: The Food Friends — The Food Friends is a research-based preschool program designed to address childhood obesity by establishing healthful eating and physical activity behaviors in preschool-aged children. The Food Friends: Fun With New Foods (12 weeks) focuses on helping children increasing children's willingness to try new foods and The Food Friends: Get Movin' With Mighty Moves (18 weeks) aims to enhance preschoolers' gross motor skill development. In effort to sustain the preschool behavior changes, the messages from The Food Friends® (Super Taster and Mighty Mover) will be extended into early elementary school through a 'booster' program. The booster program will consist of a kindergarten and 1st grade curriculum with 5 monthly units.
  Arms: Nutrition and Physical Activity

SUMMARY:
The Colorado Longitudinal Eating And Physical activity (LEAP) Study utilizes a social ecological approach to explore individual, family and environmental factors and their relationship to child weight status over a 3 year timeframe. Our primary research questions are as follows:

1. Are behavior changes (increased willingness to try new foods and gross motor skills) from a preschool nutrition and activity program, The Food Friends®, sustained through early elementary school?
2. Do The Food Friends® programs have an impact on reducing the percentage of children considered overweight and/or obese over a 3 year timeframe?
3. Do food preference and gross motor performance directly affect child weight status or are they mediators to dietary intake and physical activity?

DETAILED DESCRIPTION:
The preschool years are a critical time to begin obesity prevention efforts as they represent a time when young children establish healthy eating habits and physical activity patterns. These habits can place children at risk for obesity and are shaped by many characteristics, including individual characteristics as well as school, family and societal environmental characteristics. Predictive behaviors, or behavioral antecedents, within these environments can influence child behaviors. While many predictive behaviors have been shown to influence dietary intake, physical activity, and weight status, two potential behavioral antecedents - food preference and motor performance - need further exploration. Understanding the context in which child behavioral patterns are developed is critical to developing a model to address childhood obesity.

The Colorado LEAP project is a longitudinal cohort study utilizing a controlled quasi-experimental design in 5 rural Colorado communities. Two communities serve as intervention communities with the other 3 as matched controls. Intervention sites receive The Food Friends® nutrition and physical activity programs in preschool and 'booster' programming in kindergarten and 1st grade. Assessments are administered 4 times - twice in preschool (Fall and Spring) and once in both kindergarten and 1st grade (Spring). Observational measures with children are conducted at the school; parent/home measures are sent home and returned to school via the child; and school personnel complete school environment and policy assessments.

ELIGIBILITY:
Inclusion Criteria:

* Children enrolled in participating schools; entering kindergarten the year after recruitment

Exclusion Criteria:

* Children not entering kindergarten within one year of recruitment.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 230 (Actual)
Dates: Start 2010-09; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change in Weight Status | baseline and 2 year follow-up
  BMIz calculated from measured height and weight. Measured at baseline, post-intervention (6 months), 1 year follow-up and 2 year follow-up.

SECONDARY OUTCOMES:
Change in Tasting Preference | baseline and 2 year follow-up
  Children's willingness to try new foods and liking for foods is assessed via a preference assessment administered to each child. Measured at baseline, post-intervention (6 months), 1 year follow-up and 2 year follow-up.
Change in Dietary Intake | baseline and 2 year follow-up
  Block Food Frequency Questionnaire will be completed by parents and lunch time consumption of 2 indicator foods will be observed and weighed by research staff. Measured at baseline, post-intervention (6 months), 1 year follow-up and 2 year follow-up.
Change in Gross Motor Skills | baseline and 2 year follow-up
  The Bruininks-Oseretsky Test (BOT-2) of Motor Proficiency, Second Edition, will be used to assess gross motor development. Measured at baseline, post-intervention (6 months), 1 year follow-up and 2 year follow-up.
Change in Physical Activity | baseline and 2 year follow-up
  Measured through pedometers and accelerometers (subsample) worn by children for 6 days. Measured at baseline, post-intervention (6 months), 1 year follow-up and 2 year follow-up.

OTHER OUTCOMES:
Changes in Parental Feeding and Activity Behaviors | baseline and 2 year follow-up
  Measured via survey. Measured at baseline, post-intervention (6 months), 1 year follow-up and 2 year follow-up.
Changes in Home Environment | baseline and 2 year follow-up
  A self report survey completed by parents to measure availability of food items, physical activity items, and sedentary devices in the home. Measured at baseline, post-intervention (6 months), 1 year follow-up and 2 year follow-up.
Preschool and School Environments | baseline
  Key preschool staff will complete the Nutrition and Physical Activity Self-Assessment for Child Care (NAP SACC) instrument to identify current center nutrition and physical activity policies and practices.
  Elementary school staff will complete the School Environment and Policy Survey (SEPS), which consists of three modules designed to capture nutrition and physical activity environments, policies and programs offered in the schools.
Oral Sensory Characteristics | baseline and 2 year follow-up
  The oral sensory sensitivity scale of The Sensory Profile is administered with parents.
Self Concept | baseline and 2 year follow-up
  The Pictorial Scale of Perceived Competence and Social Acceptance for Young Children (PSPCSA) is a self-report instrument designed to assess perceptions of young children ages four to seven in four domains (i.e., Cognitive Competence, Physical Competence, Peer Acceptance, Maternal Acceptance).

CONTACTS AND LOCATIONS:
Overall Officials: Laura L Bellows, Principal Investigator — Colorado State University
Locations (6):
- United States (6):
  - Brush School District RE 2J, Brush, Colorado
  - Buena Vista School District, Buena Vista, Colorado
  - Iliff Head Start, Iliff, Colorado
  - Lake County School District, Leadville, Colorado
  - Salida School District, Salida, Colorado
  - RE-1 Valley School District, Sterling, Colorado

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Johnson SL, Ryan SM, Kroehl M, Moding KJ, Boles RE, Bellows LL. A longitudinal intervention to improve young children's liking and consumption of new foods: findings from the Colorado LEAP study. Int J Behav Nutr Phys Act. 2019 Jun 3;16(1):49. doi: 10.1186/s12966-019-0808-3. PMID 31159810
- [Derived] Boles RE, Johnson SL, Burdell A, Davies PL, Gavin WJ, Bellows LL. Home food availability and child intake among rural families identified to be at-risk for health disparities. Appetite. 2019 Mar 1;134:135-141. doi: 10.1016/j.appet.2018.12.002. Epub 2018 Dec 13. PMID 30553878
- [Derived] Johnson SL, Moding KJ, Maloney K, Bellows LL. Development of the Trying New Foods Scale: A preschooler self-assessment of willingness to try new foods. Appetite. 2018 Sep 1;128:21-31. doi: 10.1016/j.appet.2018.05.146. Epub 2018 May 26. PMID 29842966
- [Derived] Johnson SL, Davies PL, Boles RE, Gavin WJ, Bellows LL. Young Children's Food Neophobia Characteristics and Sensory Behaviors Are Related to Their Food Intake. J Nutr. 2015 Nov;145(11):2610-6. doi: 10.3945/jn.115.217299. Epub 2015 Sep 30. PMID 26423739
- [Derived] Bellows LL, Johnson SL, Davies PL, Anderson J, Gavin WJ, Boles RE. The Colorado LEAP study: rationale and design of a study to assess the short term longitudinal effectiveness of a preschool nutrition and physical activity program. BMC Public Health. 2013 Dec 9;13:1146. doi: 10.1186/1471-2458-13-1146. PMID 24321701